CLINICAL TRIAL: NCT06352060
Title: Dynamic Data-Driven Management of Atrial Fibrillation Using Implantable Cardiac Monitors: The MONITOR-AF Study
Status: Completed | Type: Observational
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: KCHRRF_MONITOR AF_030
Record Dates: First submitted 2024-02-29; First posted 2024-04-08 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with ICM: Patients who underwent ICM insertion
  Interventions: Other: No intervention or administration will be performed due to the observational nature of the study
- Non-ICM Participants: Patients with traditional monitoring methods
  Interventions: Other: No intervention or administration will be performed due to the observational nature of the study

INTERVENTIONS:
Other: No intervention or administration will be performed due to the observational nature of the study — Charts of patients enrolled in the study will be reviewed for an initial monitoring method and any changes in management.

SUMMARY:
Observational, multi-center, retrospective study to evaluate the use of ICM (implantable cardiac monitor) versus traditional, non-ICM (non-implantable cardiac monitor) methods such as ECGs (electrocardiogram), Holter, and mobile cardiac outpatient telemetry (MCOT) units.

DETAILED DESCRIPTION:
Even with its increasing popularity and use, the impact of ICMs on AF (atrial fibrillation) management is still being determined and can even be conflicting. Furthermore, the use of ICM is dependent on physician preference. It is hypothesized that dynamic monitoring with ICMs is superior to conventional methods and should be used for all patients with AF. Thus, it aimed to measure the outcomes of using ICM versus more traditional approaches in patients with AF.

ELIGIBILITY:
Inclusion Criteria

* Patients > 18 years of age
* Present for management of AF
* ICM is inserted at the discretion of the treating physician

Exclusion Criteria

* Patients < 18 years of age
* Presence of a permanent pacemaker, implantable cardiac defibrillator, or cardiac resynchronization therapy
* Unable to tolerate ICM or traditional monitoring with ECG, Holter, or MCOT monitoring
* Unable to tolerate AAD, OAC, and CA as part of AF standard of care
* ICM inserted for cryptogenic stroke or syncope
* Was not followed > 12 months
* CA performed for AF before ICM implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with atrial fibrillation management either with ICM or routine management
Sampling Method: Non-Probability Sample
Enrollment: 598 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (7):
- United States (7):
  - Menorah Medical Center, Overland Park, Kansas
  - Kansas City Heart Rhythm Institute - Roe Clinic, Overland Park, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas
  - Centerpoint Medical Center Clinic, Independence, Missouri
  - Centerpoint Medical Center, Independence, Missouri
  - Research Medical Center Clinic, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Israel CW, Gronefeld G, Ehrlich JR, Li YG, Hohnloser SH. Long-term risk of recurrent atrial fibrillation as documented by an implantable monitoring device: implications for optimal patient care. J Am Coll Cardiol. 2004 Jan 7;43(1):47-52. doi: 10.1016/j.jacc.2003.08.027. PMID 14715182
- [Background] Reiffel JA, Verma A, Kowey PR, Halperin JL, Gersh BJ, Elkind MSV, Ziegler PD, Kaplon RE, Sherfesee L, Wachter R; REVEAL AF Investigators. Rhythm monitoring strategies in patients at high risk for atrial fibrillation and stroke: A comparative analysis from the REVEAL AF study. Am Heart J. 2020 Jan;219:128-136. doi: 10.1016/j.ahj.2019.07.016. PMID 31862084
- [Background] Svendsen JH, Diederichsen SZ, Hojberg S, Krieger DW, Graff C, Kronborg C, Olesen MS, Nielsen JB, Holst AG, Brandes A, Haugan KJ, Kober L. Implantable loop recorder detection of atrial fibrillation to prevent stroke (The LOOP Study): a randomised controlled trial. Lancet. 2021 Oct 23;398(10310):1507-1516. doi: 10.1016/S0140-6736(21)01698-6. Epub 2021 Aug 29. PMID 34469766
- [Background] Reiffel JA, Verma A, Kowey PR, Halperin JL, Gersh BJ, Wachter R, Pouliot E, Ziegler PD; REVEAL AF Investigators. Incidence of Previously Undiagnosed Atrial Fibrillation Using Insertable Cardiac Monitors in a High-Risk Population: The REVEAL AF Study. JAMA Cardiol. 2017 Oct 1;2(10):1120-1127. doi: 10.1001/jamacardio.2017.3180. PMID 28842973

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 598 patients, with 299 in the non-ICM and ICM groups, respectively were included in the study.
Period: Overall Study
Arm/Group | Participants With ICM | Non-ICM Participants
Started | 299 | 299
Completed | 299 | 299
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With ICM | Non-ICM Participants | Total
Number analyzed (Participants) | 299 | 299 | 598
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.3 (7.6) | 72.3 (7.6) | 72.3 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 57 | 136
  Male | 220 | 242 | 462
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucacian | 251 | 258 | 509
  African American | 37 | 35 | 72
  Hispanic | 4 | 3 | 7
  Other | 7 | 3 | 10
Parosysmal Atrial Fibrillation [Count of Participants; unit: Participants] | 171 | 234 | 405
Persistent Atrial Fibrillation [Count of Participants; unit: Participants] | 128 | 65 | 193
Baseline AAD Use [Count of Participants; unit: Participants] | 120 | 101 | 221
Stroke / TIA [Count of Participants; unit: Participants] | 7 | 7 | 14
Compensated heart failure (EF <35%) [Count of Participants; unit: Participants] | 18 | 18 | 36
Coronary artery disease [Count of Participants; unit: Participants] | 50 | 70 | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Freedom From AF, OAC and AAD Use
Description: Number of patients with freedom from AF, OAC and AAD Use after 12 months
Time Frame: 12 Months. Data collection was 1 month examining participants retrospectively at a 1 year follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With ICM | Non-ICM Participants
Number analyzed (Participants) | 299 | 299
Participants
  Number of patients with freedom from AF | 257 | 185
  Number of patients with freedom from OAC use | 208 | 118
  Number of patients with freedom from AAD use | 230 | 109

2. Secondary Outcome: Clinical Outcomes in Participants With ICM and Non-ICM Participants
Description: Clinical Outcomes in Participants With ICM and Non-ICM Participants at 12 months
Time Frame: 12 Months. Data collection was 1 month examining participants retrospectively at a 1 year follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With ICM | Non-ICM Participants
Number analyzed (Participants) | 299 | 299
Participants
  Access to EP | 299 | 180
  Attempted Rhythm Control With AAD | 299 | 189
  OAC Compliance | 233 | 216
  Initial Ablation | 275 | 185

3. Secondary Outcome: Total CV-related Hospital Stay Duration, Days
Time Frame: 12 Months. Data collection was 1 month examining participants retrospectively at a 1 year follow-up.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Participants With ICM | Non-ICM Participants
Number analyzed (Participants) | 299 | 299
Days | 3.5 (1.9) | 7.4 (5.3)

ADVERSE EVENTS:
Time Frame: 12-Months. Data collection was 1 month examining participants retrospectively at a 1 year follow-up.
Description: All-Cause Mortality events were not monitored/assessed.
Arm/Group | Participants With ICM | Non-ICM Participants
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 7/299 | 24/299
Other Adverse Events (participants affected / at risk) | 2/299 | 9/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With ICM (N=299) | Non-ICM Participants (N=299)
AF-related hospitalization (Cardiac disorders) | 3 | 11
HF-related hospitalization (Cardiac disorders) | 4 | 13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With ICM (N=299) | Non-ICM Participants (N=299)
Stroke/TIA (Cardiac disorders) | 1 | 7
Major bleeding episodes (Blood and lymphatic system disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT06352060/Prot_SAP_000.pdf